CLINICAL TRIAL: NCT05297266
Title: Early Discovery of Ischemia After Replantation Surgery of the Extremities (EDIR-study) ; An Open, Prospective, Intervention Study
Brief Title: Early Discovery of Ischemia After Replantation Surgery of the Extremities
Acronym: EDIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sensocure AS (Industry)
Responsible Party: Principal Investigator, Magne Røkkum, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REK SØR-ØST B, ref 340841
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Ischemia; Blood Circulation Disorder; Carbon Dioxide; Biosensing Techniques; Amputation, Traumatic
Keywords: Ischemia; Biosensor; Replantation; Carbon dioxide; Traumatic amputation; Orthopedic surgery; Limb
MeSH Terms: conditions — Ischemia; Amputation, Traumatic

STUDY DESIGN:
Intervention Model Description: Prospective, interventional. Sixty patients (80 injured extremities) will receive tissue CO2 monitoring in the replanted extremity after traumatic amputation replant surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with replanted extremity monitored by tissue CO2 (Experimental): Patients with traumatic amputation of a limb who are undergoing replantation surgery and are monitored postoperatively with IscAlert biosensor measuring local tissue CO2 and temperature in the replanted extremity
  Interventions: Device: IscAlert

INTERVENTIONS:
Device: IscAlert — Insertion of a CO2- and temperature sensor in the distal part of the replanted extremity

SUMMARY:
Investigators will test if changes in CO2 is detected postoperatively in ischemic tissue in a replanted extremity of a traumatically amputated upper or lower extremity. IscAlert is measuring continuously CO2 in muscular and subcutaneous tissue. IscAlert is inserted distal to the operative field into normal muscle and/or subcutaneous tissue in the replanted extremity. Local tissue CO2 and temperature will be monitored continuously postoperatively for the next 10 days. If a reduced or totally obstructed blood flow appear (thrombosis), an increase in tissue CO2 and a lower local temperature will emerge rapidly as a sign of ischemia. This will be detected by the sensor which will alarm the investigators. This will lead to assessment of the replanted extremity and if restricted blood flow is diagnosed, a reoperation will be performed. After reoperation new sensors will be implanted for another ten days if applicable. Sixty patients will be enrolled to undergo the procedures. The IscAlert will be removed from the patient before the patient is discharged from the hospital or a maximum of 10 days (the event that occurs first). 500 devices is planned to be used in this clinical study.

DETAILED DESCRIPTION:
This is an open, prospective, interventional, single-center clinical investigation designed to examine the feasibility and safety of the IscAlert™ device in patients scheduled for extremity replant surgery. Sixty patients will be enrolled to undergo the procedures using a total of 400 devices depending on the injuries.

IscAlert is 0.8 mm in diameter and in vitro testing, shows stable and accurate measurements of pCO2. More than 200 animal experiments have been done with the sensor. The experiments have shown that the sensor detects ischemia (Increased CO2-measurements) in real time in the following organs and tissues: Brain, heart, liver, kidneys, pancreas, intestines, musculature and subcutaneous tissue. Sensitivity and specificity are close to 100%. The sensors are inserted into tissue by a split needle technique. The split needle is the size of a 3-gauge peripheral venous catheter. In animal studies, no complications have been detected when using the sensor.

The IscAlert catheters are connected to an electronics unit that is fixed to the skin with an adhesive plaster or glue outside the sterile area. The electrical signals are redirected to a PC approved for clinical use which continuously records tissue pressures of CO2.

IscAlert is inserted into normal muscle and/or subcutaneous tissue distal on the replanted limb to be operated at the end of surgery or immediate postoperatively. The insertion is far away from the operating field. The insertion is done under sterile conditions in accordance with standard sterility criteria at the hospital. No pain during insertion will occur because of insertion is performed during anesthesia (general or regional). Also, the insertion can be compared to an intramuscular injection.

Postoperatively, the IscAlert sensor will continuously monitoring tissue CO2 and temperature. If ischemia occur, for examples caused by a thrombus, an increase in tissue CO2 and a lower temperature will evolve. This will be detected by the sensor which will alarm the investigators. This will lead to assessment of the replanted extremity and if restricted blood flow is diagnosed or suspected, a reoperation will be performed.

Sixty patients will be enrolled to undergo the procedures. The IscAlert will be removed from the patient before the patient is discharged from the hospital or a maximum of 10 days (the event that occurs first). Approximately 500 devices in 80 injured extremities is planned to be used in this clinical study.

The primary objective is to compare CO2-levels in the replanted extremity in individuals who has undergone extremity replantation surgery and investigate if CO2-level is different in patient diagnosed with obstructed blood flow vs. patients with sufficient blood flow in the replanted extremity.

Our hypotheses are:

1. The IscAlert™ device will be able to detect the presence of ischemia in the extremity replant by increased pCO2 levels and decrease in tissue temperature, measured by IscAlert™.
2. By using the IscAlert™ device monitoring ischemic events, an early treatment for ischemia could lead to higher incidence of replantation survival rates, and less revision surgery caused by replantation thrombosis.
3. No clinically significant bleeding or infection will occur using IscAlert™ in this clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be in need of extremity replantation surgery
* Subject must be ≥ 18 years
* Able to give written signed informed consent

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Tissue CO2-level | 10 days
  Tissue CO2-level (kPa) during insertion period

SECONDARY OUTCOMES:
Bleeding | 10 days
  Amount of blood from insertion site (ml)
Infection | 30 days
  Infection from insertion site at the discretion of the investigator (yes or no)
Length of stay at hospital | 30 days
  Number of days from end of initial operation to primary hospital discharge + Number of days from transfer from primary hospital to discharge from secondary hospital.
Time to reduced blood flow in replanted extremity | 10 days
  Number of days and hours from primary replant surgery end to obstructed blood flow is diagnosed.
Number of re-operations | 30 days
  Number of reoperations caused by replant necrosis/ischemia in the replanted extremity

OTHER OUTCOMES:
Number of pack-years | 30 days
  Smoking habit; number of pack-years by participants
Preoperative ischemia time | 12 hours
  Preoperative ischemia time of the amputated limb (minutes)
Intravenous fluid | 12 hours
  Intravenous fluid given during surgery (ml)
Vasoactive drugs | 10 hours
  Vasoactive drugs given during surgery (microgram)
IscAlert functionality | 10 days
  Number of hours with a well-functioning sensor (giving CO2- and temperature data)
Physical examination of the reimplanted extremity - capillary filling | 10 days
  Time of capillary filling (seconds)
Physical examination of the reimplanted extremity - color | 10 days
  Color of reimplanted extremity (Red or Pale)
Physical examination of the reimplanted extremity - temperature | 10 days
  Temperature of reimplanted extremity (degrees Celsius)

CONTACTS AND LOCATIONS:
Overall Officials: Magne Røkkum, MD, Ph.D, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD to other researchers